CLINICAL TRIAL: NCT04294433
Title: Clinical Trial to Assess Immunogenicity of 2 Versus 3 Doses of Hepatitis B Vaccines When Administered to Children Aged 2 to 18 Months
Brief Title: Immunogenicity of 2 Versus 3 Doses of Combined Hepatitis B Vaccines in 2-18 Months Old Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Study 11022017
Record Dates: First submitted 2020-01-29; First posted 2020-03-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis B
Keywords: Vaccination; Two doses; Infants; Clinical trial; Hepatitis B; Heterologous schedule; Immunogenicity; Randomization; Reduced-dose schedule
MeSH Terms: conditions — Hepatitis B | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Intervention Model Description: Randomised 1:1 for 2 study groups. Non-randomised for comparator group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infanrix-hexa+Infanrix-hexa+Infanrix-hexa (Active Comparator): Children vaccinated at the age of 2, 4 and 18 months with a standard dose of Infanrix-hexa
  Interventions: Biological: Infanrix-hexa
- Infanrix-hexa+Infanrix-hexa (Experimental): Children vaccinated at the age of 2 and 12 months with a standard dose of Infanrix-hexa
  Interventions: Biological: Infanrix-hexa
- Infanrix-hexa+Twinrix Junior (Experimental): Children vaccinated at the age of 2 and 12 months with a standard dose of Infanrix-hexa and a standard dose of Infanrix-Junior, respectively
  Interventions: Biological: Infanrix-hexa and Twinrix Junior

INTERVENTIONS:
Biological: Infanrix-hexa — Vaccines administrated according to product monographs' recommendations
  Arms: Infanrix-hexa+Infanrix-hexa; Infanrix-hexa+Infanrix-hexa+Infanrix-hexa
Biological: Infanrix-hexa and Twinrix Junior — Vaccines administrated according to product monographs' recommendations
  Arms: Infanrix-hexa+Twinrix Junior

SUMMARY:
The main objective of this study is to compare the immunogenicity of the hepatitis B component in children vaccinated with (I) two doses of Infanrix-hexa administered at 2 and 12 months of age versus (II) one dose of Infanrix-hexa and one dose of Twinrix administered respectively at 2 and 12 months of age versus (III) three doses of Infanrix-hexa administered at 2, 4 and 18 months of age (comparator).

DETAILED DESCRIPTION:
In the province of Quebec, Canada, hepatitis B vaccination of infants involves three doses of vaccine, 2, 4 and 18 months of age. However, in the current epidemiological context (virtual absence of new cases in young Quebecers) and taking into account scientific data which consistently show a high immunogenicity and efficacy of two doses of hepatitis B vaccine, the relevance of the second dose given at the age of 4 months is questionable.

this study is designed to compare the immunogenicity of the hepatitis B component in children vaccinated with (I) two doses of Infanrix-hexa administered at 2 and 12 months of age versus (II) one dose of Infanrix-hexa and one dose of Twinrix administered respectively at 2 and 12 months of age versus (III) three doses of Infanrix-hexa administered at 2, 4 and 18 months of age (comparator).

ELIGIBILITY:
Inclusion Criteria:

* Comparator group :
* Have received 3 doses of Infanrix-hexa as part of the regular vaccination program at the age of 2, 4 and 18 months.
* Study groups:
* Have received 1 dose of Infanrix-hexa as part of the regular vaccination program at the age of 2 months.

Exclusion Criteria:

* Have received other doses of hepatitis B vaccine;
* Considered immunosuppressed;
* Have an autoimmune disease;
* Have contraindications to HBV vaccination, as defined in the Quebec Immunization Protocol;
* Have a bleeding disorder;

  * Have a significant developmental delay;
  * Have or plan to participate in other clinical studies with vaccines or products not licensed in Canada;
  * Have presented a serious clinical condition to the vaccines administered as part of the study.

Ages: 2 Months to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 431 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Immunogenicity - Seroprotection | 1 month after the primary series
  The proportion of children with an anti-HBs titer ≥10mIU/ml
Immune memory - Anamnestic response | 1 month after a challenge dose administered 36 months after the end of the primary series
  Immune response to a challenge dose: anti-HBs titers at least 10 mIU/mL and a fourfold increase in titers

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Laval University Research Hospital Center, Québec, Quebec
  - Équipe de recherche en vaccination, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared with any other researchers outside of this study